CLINICAL TRIAL: NCT05758311
Title: Adipose Tissue & Adipokines (ATA): From Laboratory to Clinical Practice - The Project ATA
Brief Title: The Project ATA: Adipose Tissue & Adipokines
Acronym: ATA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dynamical Business and Science Society - DBSS International SAS (Network)
Collaborators: CES University (Other); Universidad de Córdoba (Other)
Responsible Party: Sponsor
Other Study IDs: ATA_DBSS
Record Dates: First submitted 2023-02-06; First posted 2023-03-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Sedentary Behavior; Overweight; Obesity
Keywords: Body Composition; Body Fat Distribution; Biomarkers; Cardiovascular Risk; Anthropometry; Bioelectrical Impedance; Adipomyokines
MeSH Terms: conditions — Sedentary Behavior; Overweight; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood samples will be collected from the forearm veins of the participants to quantify the concentration of adipokines and lipid profile.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multi-center study: The study population will be inhabitants of both sexes with different levels of physical activity who reside in the metropolitan area of cities in Colombia, Mexico, Costa Rica, and Spain. The population sample will be obtained through an internal call to students and administrative personnel of universities and Smart Fit sites with an inter-institutional collaboration agreement with Dynamical Business & Science Society (DBSS International). The first study will be carried out in Colombia.

SUMMARY:
It is essential to delve deeper into the molecular and tissue aspects that allow us to recognize the roles of adipose tissue and its interaction with the musculoskeletal (i.e., adipomyokines) to facilitate the identification of biomarkers that can complement the assessment of body composition. Thus, investigators posed the following research question: what characteristics of adipose tissue can investigators consider to rethink assessment for the diagnosis and treatment of obesity? The 'Project ATA' is a cross-sectional study based on the Strengthening the Reporting of Observational Studies in Epidemiology-Nutritional Epidemiology (STROBE-nut) guidelines, an Extension of the STROBE Statement. The FINER strategy (Feasible, Interesting, Novel, Ethical, and Relevant) and previously published guidelines for organizing a multicenter study will be followed. The 'Project ATA' will test the associations of several morphological metrics and adipomyokines in order to both profile populations with excess body fat and to establish practical geographical-based recommendations for practitioners.

DETAILED DESCRIPTION:
Obesity is a multifactorial disease characterized by excess and accumulation of body fat, which implies hypertrophy and hyperplasia of adipocytes (i.e. adipose tissue cells). However, obesity is not only related to lipid accumulation in adipose tissue but could also generate morpho-functional changes in other tissues. The deleterious effects of lipid accumulation in non-adipose tissues are known as lipotoxicity. Lipotoxicity generates certain metabolic alterations, which affect overall metabolic health, leading to ectopic fat accumulation (i.e. fat accumulation outside its proper place). These factors can result in an increased likelihood of chronic diseases, including cardiovascular disease, type 2 diabetes mellitus, non-alcoholic fatty liver disease, chronic kidney disease, and different types of cancer. There is substantial variation between individuals, some obese people may remain metabolically healthy and some lean people may have metabolic diseases. Additionally, adipose tissue in addition to having an energy storage role produces hormones that regulate different physiological processes, such as inflammatory responses, mechanical cushioning and insulation, and participation in heat production for body temperature regulation. These processes can change adaptively (or maladaptation) during the loss or gain of body mass. Importantly, insufficient adipose tissue (lipodystrophy) or adipose tissue dysfunction (e.g. obesity) leads to excessive lipid deposition in other organs such as the liver and muscle.

Obesity comprises much damage in different tissues of the organism; however, these changes are potentially reversible by taking advantage of the innate property of biological systems to favor adaptation to repeated stimuli (e.g., changes in habits and lifestyles). The particularity of obesity is the expansion of adipose tissue, although this does not always mean that it is pathological. A clear example is natural obesity in various mammals during the pre-hibernation stage and subsequent periods of high physical activity. Healthy adipose tissue expansion is accompanied by adequate capillary angiogenesis and mitochondria-centered metabolic control. On the other hand, unhealthy adipose tissue expansion is associated with capillary and mitochondrial impairment, resulting in immune cell deposition and excessive production of proinflammatory cytokines. In addition, some pathologies of metabolically healthy obese individuals have well-preserved adipose tissue function, associated with fewer comorbidities and lower mortality rates compared to lean individuals.

The reasons for studying beyond the energetic function of adipose tissue are based on the plasticity of adipose tissue and its different types (both morphological and metabolic). Traditionally, adipose tissue is classified as white adipose tissue (WAT), brown adipose tissue (BAT), and beige adipose tissue (bAT). However, other types of adipose tissue have been identified, including pink and yellow (bone marrow) adipose tissue, highlighting their physiological functions after trans-differentiation processes. It is necessary to establish an understanding of the complexity of adipose tissue and its endocrine interaction with other tissues to determine the physiological response to external stimuli (e.g., overenergetic diet, physical inactivity, sedentary lifestyle, cancer, etc.). In fact, a geographical variation of obesity and the associated risk factors has been reported by different research groups. This questions and highlights the need to improve the obesity metrics for diagnosis and monitoring.

The aim of 'Project ATA' is double: i) to profile the population with excess fat mass (overweight and obesity) using body composition data and the concentration of adipomyokines, and ii) to evaluate the association between morphophysiological and endocrine variables in order to propose practical geographical-based recommendations to assess and monitor obesity accurately.

ELIGIBILITY:
Inclusion Criteria:

* People over 18 years of age (under 60 years of age).
* People born and residing in major cities or neighboring municipalities of the metropolitan area of selected cities. The first stage will take place in Medellín (Colombia) and then continue in other cities in Colombia, Costa Rica, Mexico, and Spain according to logistics procedures.
* Those who sign the informed consent to undergo the measurements.

Exclusion Criteria:

* Those physically active people who exercise vigorously and systematically or at a competitive level.
* Those diagnosed with a musculoskeletal disease and/or special condition that limits mobility during the taking of measurements (musculoskeletal injury).
* People over 60 years of age.
* Pregnant women.
* People with implants or synthetic prostheses.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be inhabitants of both sexes with different levels of physical activity who reside in the metropolitan area of cities in Colombia, Mexico, Costa Rica, and Spain. Investigators will primarily consider university students, administrative personnel, and other potentially eligible adults of both sexes who respond to the study announcement, fulfill inclusion criteria and sign the informed consent form. To understand the prevalence or proportion of a given phenotype among adults in a city a formula based on previously reported proportions will be used to calculate the sample size.
Sampling Method: Non-Probability Sample
Enrollment: 378 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Anthropometric Assessment | July 2023 to August 2024
  All measurements will be performed according to the International Standards for Anthropometric Evaluation published by the International Society for the Advancement of Kineanthropometry (ISAK) to obtain basic measurements expressed in absolute data. Means will be calculated and analyzed from two measurements of anthropometric data.
Anthropometry-Based Analysis of Body Composition | July 2023 to August 2024
  The whole-body fat percentage (RFM), the sum of skinfolds, the waist girth (minimal and umbilicus), the body mass to waist girth, waist girth to stature ratios. Finally, musculoskeletal index, the skinfold-corrected muscle girths for the arm, chest, waist, thigh, and calf will be calculated according to the expression: girth - (π x skinfold).
Bioelectrical Impedance Analysis | July 2023 to August 2024
  To evaluate adult subjects with excess adiposity by foot-to-foot bioelectrical impedance analysis (BIA). Estimated values of percent fat mass (FM), percent muscle mass (MA), metabolic age (ma), basal metabolic rate (BMR), and visceral fat (VFL). In addition, bioelectrical impedance vector analysis (BIVA) will be performed and raw variables related to phase angle and body composition will be reported.
Adipokines and blood screening | July 2023 to August 2024
  Will be collected peripheral blood samples, where it will be taken into account serum amyloid A, resistin, leptin, adiponectin, and visfatin concentrations will be quantified by direct chemiluminescence using acridinium ester technology.

CONTACTS AND LOCATIONS:
Overall Officials: Diego A Bonilla, MSc, Principal Investigator — Research Division, Dynamical Business & Science Society - DBSS International SAS, Bogotá, Colombia; Luis M Gómez-Miranda, PhD, Principal Investigator — Sports School, Autonomous University of Baja California, Tijuana 22390, México; Daniel Rojas-Valverde, PhD, Principal Investigator — Núcleo de Estudios para el Alto Rendimiento y la Salud (CIDISAD-NARS), Heredia, Costa Rica; Salvador Vargas-Molina, MSc, Principal Investigator — Faculty of Sport Sciences, EADE-University of Wales Trinity Saint David, 29018 Málaga, Spain; Katherine Franco-Hoyos, MSc, Principal Investigator — Nutral, Universidad CES, Medellín, Colombia
Locations (1):
- DBSS, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No
The data collected in this study will be used for research purposes, according to the bioethical standards established by the Institutional Review Board (IRB) and the procedures will be developed in accordance with the latest version of the Declaration of Helsinki. Investigators will not share the identity of those who participate in the research. The information investigators collect in this research project will be kept confidential, will be kept off-limits, and no one except the researchers will have access to it. Any information about the participant will have an identifying number (rather than the name) at the time of analysis. Only the researchers will know what the number is and the information will be kept confidential. It will not be shared or given to anyone except participants, a Data and Safety Monitoring Board (DSMB), or others participants authorize (e.g., physician, nutritionist).

REFERENCES:
- [Background] Apovian CM. Obesity: definition, comorbidities, causes, and burden. Am J Manag Care. 2016 Jun;22(7 Suppl):s176-85. PMID 27356115
- [Background] Bonilla DA, De Leon LG, Alexander-Cortez P, Odriozola-Martinez A, Herrera-Amante CA, Vargas-Molina S, Petro JL. Simple anthropometry-based calculations to monitor body composition in athletes: Scoping review and reference values. Nutr Health. 2022 Mar;28(1):95-109. doi: 10.1177/02601060211002941. Epub 2021 Apr 1. PMID 33792415
- [Background] Bremner JD, Moazzami K, Wittbrodt MT, Nye JA, Lima BB, Gillespie CF, Rapaport MH, Pearce BD, Shah AJ, Vaccarino V. Diet, Stress and Mental Health. Nutrients. 2020 Aug 13;12(8):2428. doi: 10.3390/nu12082428. PMID 32823562